CLINICAL TRIAL: NCT06871631
Title: Relationships Between Serum Vitamin D Levels and Osteocalcin and N-terminal Telopeptide Levels in Gingival Crevicular Fluid
Brief Title: Serum Vitamin D and Gingival Crevicular Fluid Levels of Osteocalcin and N-Terminal Telopeptide
Status: Completed | Type: Observational
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Atanur Sarioglu, Research assistant, Ondokuz Mayıs University
Other Study IDs: OMU KAEK protokol no: 2017/60
Record Dates: First submitted 2025-03-04; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: D Vitamin Deficiency; Osteocalcin; Gingival Crevicular Fluid
Keywords: Vitamin D; Osteocalcin; N-Terminal Telopeptide; Gingival Crevicular Fluid
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- Patients with periodontitis and 25(OH)D levels of 0-10 ng/ml: Patients diagnosed with periodontitis who have serum 25-hydroxyvitamin D [25(OH)D] levels ranging from 0 to 10 ng/ml.
- Patients with periodontitis and 25(OH)D levels of 11-20 ng/ml: Patients diagnosed with periodontitis who have serum 25-hydroxyvitamin D [25(OH)D] levels ranging from 11 to 20 ng/ml.
- Patients with periodontitis and 25(OH)D levels of 21-30 ng/ml: Patients diagnosed with periodontitis who have serum 25-hydroxyvitamin D [25(OH)D] levels ranging from 21 to 30 ng/ml.
- Periodontally healthy patients and 25(OH)D levels of 0-10 ng/ml: Periodontally healthy patients with serum 25-hydroxyvitamin D [25(OH)D] levels between 0 and 10 ng/ml.
- Periodontally healthy patients and 25(OH)D levels of 11-20 ng/ml: Periodontally healthy patients with serum 25-hydroxyvitamin D [25(OH)D] levels between 11 and 20 ng/ml.
- Periodontally healthy patients and 25(OH)D levels of 21-30 ng/ml: Periodontally healthy patients with serum 25-hydroxyvitamin D [25(OH)D] levels between 21 and 30 ng/ml.

SUMMARY:
This study examines the relationship between serum vitamin D levels and bone metabolism markers-osteocalcin and N-terminal telopeptide (NTx)-in gingival crevicular fluid (GCF) of periodontally healthy and periodontitis patients. A total of 120 male participants (60 healthy, 60 with periodontitis) aged 25-40 were included and categorized based on their serum vitamin D levels.

DETAILED DESCRIPTION:
Recent evidence suggests that vitamin D, a key regulator of bone metabolism, may play a role in periodontal health by influencing bone turnover markers such as osteocalcin and N-terminal telopeptide (NTx). This study aims to investigate the effects of serum vitamin D levels on these bone metabolism markers in gingival crevicular fluid (GCF) of periodontally healthy and periodontitis patients.

A total of 120 male participants aged 25-40 years were enrolled, comprising 60 periodontally healthy individuals and 60 patients diagnosed with periodontitis. Participants were further categorized into subgroups based on their serum vitamin D levels (0-10 ng/ml, 11-20 ng/ml, and 21-30 ng/ml). GCF samples were collected from maxillary premolar and molar sites and analyzed using enzyme-linked immunosorbent assay (ELISA) to measure osteocalcin and NTx concentrations.

ELIGIBILITY:
Inclusion Criteria:

* One hundred and twenty male patients, consisting of 60 periodontally healthy patients and 60 patients with periodontitis, aged between 25 and 40 years, non-smoking, who had not received periodontal treatment in the last 6 months, with no systemic diseases, and whose Vitamin D levels had been determined, were included in the study.

Exclusion Criteria:

* Female individuals
* Smokers
* Individuals with systemic diseases (Diabetes Mellitus, Hyperthyroidism, -Malabsorption, Liver and Renal Failure, or those receiving osteoporosis treatment)
* Individuals who have undergone periodontal treatment within the last 6 months
* Individuals on regular medication
* Individuals who did not provide informed consent
* Individuals with poor cooperation

Ages: 25 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — One hundred and twenty male patients, consisting of 60 periodontally healthy patients and 60 patients with periodontitis, aged between 25 and 40 years.
Study Population: Study participants will be selected from individuals seeking care at the Department of Periodontology, Faculty of Dentistry, and the Department of Endocrinology, Faculty of Medicine, Ondokuz Mayis University, Samsun, Turkey. The population includes adults with varying periodontal and vitamin D statuses, including periodontally healthy individuals and those with periodontitis. Participants represent a diverse clinical population from the surrounding region and are recruited based on their eligibility for the study's objectives, particularly in relation to serum vitamin D levels and bone metabolism markers in gingival crevicular fluid.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2018-06-10 (Actual); Primary Completion 2022-04-17 (Actual); Study Completion 2025-02-15 (Actual)

PRIMARY OUTCOMES:
Osteocalcin Concentration in Gingival Crevicular Fluid (ng/mL) | At baseline (single time point)
  Osteocalcin concentration will be determined using an enzyme-linked immunosorbent assay (ELISA) and expressed in ng/mL.
N-Terminal Telopeptide Concentration in Gingival Crevicular Fluid (nmol/L) | At baseline (single time point)
  NTx concentration will be measured using an ELISA and expressed in nmol/L.
Total Osteocalcin Levels in Gingival Crevicular Fluid (ng/ml) | At baseline (single time point)
  This measure assesses the total osteocalcin amount in gingival crevicular fluid. Absorbance values will be recorded using an ELISA reader, and total levels will be determined based on a standard curve.
Total N-Terminal Telopeptide Levels in Gingival Crevicular Fluid (nmol/L) | At baseline (single time point)
  This measure quantifies the total amount of N-Terminal Telopeptide in gingival crevicular fluid. The total amount is determined using ELISA and calculated based on a standard curve.

SECONDARY OUTCOMES:
Corelation between serum vitamin D levels (ng/ml) and osteocalcin (ng/ml) and N-terminal telopeptide levels (nmol/L) in gingival crevicular fluid | At baseline (single time point)
  This outcome measure evaluates the correlation between serum vitamin D levels and osteocalcin and N-terminal telopeptide levels in gingival crevicular fluid across different vitamin D ranges and periodontal health statuses. Serum vitamin D levels will be categorized into three groups: 0-10 ng/mL, 11-20 ng/mL, and 21-30 ng/mL. Participants will be classified as periodontally healthy or having periodontitis based on clinical periodontal assessments.
Periodontal clinical parameters (probing depth) | At baseline (single time point)
  Probing depth of ≤3 mm was recorded as within the normal healthy range, while ≥5 mm was considered unhealthy
Periodontal clinical parameters (bleeding on probing) | At baseline (single time point)
  Bleeding on probing (BoP) <10% was considered within the healthy range, while ≥10% was classified as unhealthy.
Periodontal clinical parameters (clinical attachment level) | At baseline (single time point)
  Clinical attachment level (CAL) was assessed based on probing depth (PD) and gingival recession, with measurements taken from the cementoenamel junction (CEJ) to the base of the pocket. Radiographic bone loss was also evaluated to confirm attachment loss and periodontal status.

CONTACTS AND LOCATIONS:
Overall Officials: Atanur Sarioglu, DDS, Principal Investigator — Ondokuz Mayıs University, Department of Periodontology
Locations (1):
- Department of Periodontology, Faculty of Dentistry, Ondokuz Mayis University, Samsun, Atakum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The decision to not share individual participant data (IPD) is based on ethical considerations, institutional policies, and the need to protect participant privacy and confidentiality. The collected data will only be used for the purposes of this study and will not be made available for external use.